CLINICAL TRIAL: NCT06108596
Title: Evaluation of the Efficacy and Safety of Interleucin-2 Combined With PD-1 Monoclonal Antibody and CAPOX in Preoperative Neoadjuvant Therapy for Mid-low Locally Advanced Rectal Cancer
Brief Title: Evaluation of the Efficacy and Safety of Interleucin-2 Combined With PD-1 Monoclonal Antibody and CAPOX in Preoperative Neoadjuvant Therapy for Mid-low Locally Advanced Rectal Cancer - a Single-center, Single-arm, Open-label Clinical Trail
Acronym: PICS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRSYM202310
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2025-01

CONDITIONS: Locally Advanced Rectal Adenocarcinoma
Keywords: Immunotherapy treatment; IL-2; Rectal cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental group (Experimental): Sintilimab with Interleukin-2+CAPOX
  Interventions: Drug: Sintilimab with Interleukin-2+CAPOX

INTERVENTIONS:
Drug: Sintilimab with Interleukin-2+CAPOX — Sintilimab with Interleukin-2+CAPOX

SUMMARY:
Evaluation of the efficacy and safety of interleucin-2 combined with PD-1 monoclonal antibody and CAPOX in preoperative neoadjuvant therapy for mid-lower locally advanced rectal cancer - a single-center, single-arm, open-label clinical trail.

DETAILED DESCRIPTION:
The global incidence rate of rectal cancer is approximately 732,000 cases/year, of which a significant proportion is locally advanced rectal cancer (i.e., T3-4 or N+). Currently, for locally advanced rectal cancer, the NCCN guidelines recommend treatment with neoadjuvant radiotherapy and chemotherapy + total mesorectal excision + adjuvant chemotherapy, reducing the local recurrence rate of locally advanced rectal cancer from over 30% to less than 10%. However, this treatment mode still has a low overall sphincter preservation rate, a high distant metastasis rate, and limited overall survival (OS) benefits. In recent years, the emergence of total neoadjuvant therapy (TNT) strategies, including induction chemotherapy + concurrent chemoradiotherapy + surgery, concurrent chemoradiotherapy + consolidation chemotherapy (two or even three drugs) + surgery, and concurrent chemoradiotherapy + consolidation immunotherapy combined with chemotherapy + surgery, have all improved the long-term prognosis of locally advanced rectal cancer to varying degrees. However, the TNT mode is not suitable for all rectal cancer patients. For patients with low or moderate-risk rectal cancer or those who cannot tolerate intensive radiotherapy and chemotherapy, TNT increases the potential risk of overtreatment and associated toxicity.

The emergence of immunotherapy, including adoptive cell transfer (ACT) and immune checkpoint inhibitors (ICB), provides new insights into the treatment of locally advanced rectal cancer. However, most colorectal cancer patients have a limited response to immunotherapy. For ACT, many clinical studies report that exogenously infused antitumor T cells have poor tumor tissue infiltration, resulting in extremely limited immune responses. This inefficiency in T cell delivery may be due to high interstitial fluid pressure, pathological vascular networks, tumor-associated fibroblasts, or the "physical barrier" of the extracellular matrix (ECM), as well as the immunosuppressive tumor microenvironment. As for immune checkpoint inhibitors (ICIs), especially PD-1/PD-L1 targeted therapies, they have shown significant promise in the treatment of various solid tumors, including breast cancer, lung cancer, gastric cancer, and colorectal cancer. Studies such as CheckMate-142 and KEYNOTE-177 have confirmed the excellent efficacy of PD-1/PD-L1 inhibitors in the treatment of colorectal cancers with mismatch repair protein defects (dMMR) or high microsatellite instability (MSI-H). Institutions like the Memorial Sloan Kettering Cancer Center (MSKCC), Sun Yat-sen University Cancer Center, and the Sixth Affiliated Hospital of Sun Yat-sen University have conducted research on PD-1 inhibitors for neoadjuvant treatment of locally advanced rectal cancer, with complete remission rates as high as 75% to 100%. However, this patient population is very small, accounting for about 15% of early-stage colorectal cancers and only 5% of advanced colorectal cancers, especially less than 5% in rectal cancer. Meanwhile, microsatellite stable (MSS) patients make up the vast majority of colorectal cancers, and they benefit little from single-agent immunotherapy.

In this population, low tumor mutation burden (TMB) and insufficient immunogenicity, leading to inadequate immune cell infiltration, are considered one of the main resistance mechanisms to immunotherapy. Therefore, enhancing immune cell infiltration and boosting the therapeutic effect of immunotherapy in low-responsive colorectal cancer has significant clinical importance. Currently, some clinical experiments are being conducted in this area. For instance, radiotherapy theoretically synergizes with immunotherapy, possibly through the release of tumor antigens, remodeling of the immune microenvironment, and increasing antitumor immune responses, thus producing a combined therapeutic effect. Prospective phase II studies suggest that radiotherapy combined with immunotherapy achieves a higher pCR rate in pMMR/MSS locally advanced rectal cancer. Additionally, various immune cells in the tumor microenvironment (TME) can impair tumor immune responses, leading to tumor resistance to PD-1 therapy. Much evidence suggests that T cells in or near tumor tissues, although activated, cannot attack tumor cells. Thus, enhancing T cell tumor infiltration and activating their antitumor effects are key methods to enhance PD-1 therapy. Recent basic research results show that elevated levels of TGF-β and VEGF in tumor tissues suppress the aforementioned cytokines, enhancing tumor T cell infiltration and the efficacy of anti-PD-1 therapy. Moreover, a phase Ib clinical trial from Australia suggests that Pixatimod (a TLR9 agonist) combined with Nivolumab shows tolerability and clinical benefits in MSS mCRC patients, and researchers also observed pharmacodynamic changes and biomarker signals related to clinical benefits in the combination scheme. Similarly, another phase I clinical trial suggests that low molecular weight heparin (LMWH) enhances the efficacy of anti-PD-1 in MSS colorectal cancer by increasing CD8+T cell infiltration. These results highlight the immense prospects of PD-1 therapy combined with immune enhancement in antitumor immunotherapy.

IL-2 (Interleukin-2) is an essential cytokine, primarily produced by activated T cells. It plays a pivotal role in the immune system by promoting the growth and differentiation of T cells, enhancing the activity of cytotoxic T cells (CTLs) and natural killer cells (NK cells), and participating in immune responses against pathogens and tumors. In past tumor treatments, the primary application of IL-2 was to initiate and amplify the body's immune attack on tumors. In the treatment of certain diseases, such as malignant melanoma and renal cancer, monotherapy with appropriate doses of IL-2 has proven beneficial. For instance, a low dose of IL-2 20IU subcutaneous injection can induce immune activation while producing fewer clinical side effects. However, the complications of high-dose IL-2 treatment can be severe, including hypotension, respiratory distress, and renal impairment. Although IL-2 has some application in tumor immunotherapy, its efficacy is often limited, benefiting only a minority of patients. Current research is exploring ways to enhance the effectiveness of IL-2, including the development of novel IL-2 variants that improve the molecule's selectivity and stability, as well as combination therapies with other immune modulators, such as checkpoint inhibitors. In certain conditions, such as Lymphocytic Choriomeningitis Virus (LCMV) infection, the combined treatment of PD-1 and IL-2 has shown remarkable clinical efficacy. In vivo experiments indicate that, compared to PD-1 monotherapy, the combination of PD-1+IL-2 for LCMV significantly alters the differentiation program of PD-1+TCF1+ stem-like CD8+T cells, producing effector CD8+T cells distinct at the transcriptional and epigenetic levels, very similar to those observed after acute viral infections. Furthermore, in head and neck squamous cell carcinoma (HNSCC), a bispecific immune cytokine PD1-IL2v can notably activate immune cells, including NK cells and CD8+T cells, and inhibit the proliferation and metastasis of tumor cells. These discovered mechanisms elucidate the potential synergy between IL-2 treatment and PD-1 blockade, providing guidance and a theoretical foundation for our clinical trial using the combination of PD-1 and IL-2 in patients with locally advanced rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged between 18 and 75 years;
2. ECOG performance status score of 0 or 1;
3. Histologically confirmed rectal adenocarcinoma;
4. Clinical stage T3-T4 or any T with positive lymph nodes (N+): locally advanced;
5. Microsatellite stable (MSS) or deficient mismatch repair (dMMR) status;
6. Distance from the anal verge ≤ 12 cm;
7. Adequate hematologic, hepatic, and renal function.

Exclusion Criteria:

1. Metastatic disease (Stage IV); recurrent colorectal cancer with active bleeding, perforation, or complex conditions requiring urgent surgery; or concurrent presence of other non-colorectal malignancies;
2. Patients who have previously received systemic anticancer therapy for colorectal cancer; or patients treated with PD-1, PD-L1, or CTLA-4 antibodies;
3. Patients with any active autoimmune disease; known or tested positive for Human Immunodeficiency Virus (HIV) or Acquired Immunodeficiency Syndrome (AIDS); or a history of treatment with steroids or immunosuppressive drugs;
4. Rectal or colon cancer located more than 12 cm from the anal verge;
5. Patients with interstitial lung disease, non-infectious pneumonia, or uncontrolled systemic diseases (e.g., diabetes, hypertension, pulmonary fibrosis, and acute pneumonia);
6. Patients who experienced any Grade 2 or higher toxicity due to previous treatments (according to Common Terminology Criteria for Adverse Events (CTCAE) version 5), which has not resolved (excluding anemia, alopecia, and skin pigmentation changes); known or suspected allergy to any of the related drugs used in the trial;
7. Pregnant or breastfeeding women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-10-21 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
pCR | From the start of initial medication to the final determination via pathology results after surgical treatment, the assessment period will be up to a maximum of 6 months.
  To evaluate whether neoadjuvant Sintilimab with Interleukin-2+CAPOX would significantly improve the pathological complete response (pCR) proportion in patients with locally advanced rectal cancer

SECONDARY OUTCOMES:
cCR | From the start of initial medication to the end of six cycles of treatment, with final determination based on radiological examination, endoscopic examination results, and other assessments, the assessment period will be up to a maximum of 6 months.
  To evaluate whether neoadjuvant Sintilimab with Interleukin-2+CAPOX would significantly improve the Clinical complete response (cCR) proportion in patients with locally advanced rectal cancer
R0 resection rate R0 resection rate | From the start of initial medication to the final determination via pathology results after surgical treatment, the assessment period will be up to a maximum of 6 months.
Major pathological response (MPR) | From the start of initial medication to the final determination via pathology results after surgical treatment, the assessment period will be up to a maximum of 6 months.
Adverse Event | From the start of initial medication to the end of six cycles of treatment, the assessment period will be up to 1 month after the last treatment.
Complications within 30 days post-surgery | within 30 days post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yueming Sun, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Jiangsu Province Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No